CLINICAL TRIAL: NCT00665561
Title: AN INTERNATIONAL, MULTICENTER, PROSPECTIVE OBSERVATIONAL STUDY OF THE SAFETY OF MARAVIROC USED WITH OPTIMIZED BACKGROUND THERAPY IN TREATMENT-EXPERIENCED HIV-1 INFECTED PATIENTS
Brief Title: Prospective Observational Epidemiologic Study of Maraviroc's Safety
Acronym: POEM
Status: Completed | Type: Observational
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A4001067; 2007-006148-24 (EudraCT Number); POEM (Other: Alias Study Number)
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Human Immunodeficiency Virus
Keywords: Maraviroc; HIV-1; Safety; Non-interventional
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Maraviroc

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Maraviroc exposed
  Interventions: Drug: Maraviroc along with an optimized background antiretroviral drug regimen
- Maraviroc unexposed
  Interventions: Drug: Optimized background antiretroviral drug regimen without maraviroc

INTERVENTIONS:
Drug: Maraviroc along with an optimized background antiretroviral drug regimen — Maraviroc prescribed per approved local label.
  Other Names: Selzentry, Celsentri
  Groups: Maraviroc exposed
Drug: Optimized background antiretroviral drug regimen without maraviroc — Optimized background antiretroviral therapy prescribed per approved local label and treatment guidelines.
  Groups: Maraviroc unexposed

SUMMARY:
The study will assess if use of maraviroc along with an optimized background regimen of antiretroviral drugs in usual clinical practice is as safe as using only an optimized regimen of antiretroviral drugs.

DETAILED DESCRIPTION:
All patients meeting the study eligibility criteria at participating sites will be invited to participate.

ELIGIBILITY:
Inclusion Criteria:

* Treatment experienced, HIV-1 infected patients
* 18 years or older
* Receive an approved assay for determination of HIV-1 tropism

Exclusion Criteria:

* Pregnant or lactating
* Using CCR5 inhibitor other than maraviroc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment experienced, HIV-1 infected patients in routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2008-03-31 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (267):
- United States (143):
  - Health Services Center, Hobson City, Alabama
  - AAC/Davis Clinic, Huntsville, Alabama
  - Alabama Infectious Diseases Center, Huntsville, Alabama
  - Office of Franco Antonio Felizarta MD, Bakersfield, California
  - Providence Clinical Research, Burbank, California
  - Lalla-Reddy Medical Corporation, Fountain Valley, California
  - Bickerstaff Pediatric Family HIV Center, Long Beach, California
  - LA Gay and Lesbian Center, Los Angeles, California
  - Office of Peter J. Ruane, MD, Los Angeles, California
  - Cedars Sinai Medical Group, Los Angeles, California
  - Alta Bates Summit Medical Center East Bay AIDS Center, Oakland, California
  - University of California Irvine Medical Center, Orange, California
  - A Professional Corporation, Research Department, Palm Desert, California
  - Stanford ACTG, Palo Alto, California
  - University of California, Sacramento, California
  - Kaiser Permanente Medical Center, San Francisco, California
  - San Francisco Veterans Affairs Medical Center, San Francisco, California
  - Statnford University Medical Center, Stanford, California
  - Bipin Bhagat MD Inc., Victorville, California
  - Kaiser Permanente, Denver, Colorado
  - National Jewish Health, Denver, Colorado
  - Kaiser Permanete of Colorado Rock Creek Medical Offices, Lafayette, Colorado
  - Yale University School of Medicine Aids Program, New Haven, Connecticut
  - Clinical AIDS & HIV, New Haven, Connecticut
  - Hospital of Saint Raphael, New Haven, Connecticut
  - Circle Medical, LLC, Norwalk, Connecticut
  - Dupont Circle Physician's Group, Washington D.C., District of Columbia
  - Family Medical Counseling Service, Washington D.C., District of Columbia
  - Division of Infectious Diseases, George Washington University Medical Center, Washington D.C., District of Columbia
  - George Washington University Medical Faculty Assoc, Washington D.C., District of Columbia
  - Office of Mahmoud H. Mustafa, MD, FACP, Washington D.C., District of Columbia
  - ID Consultants Inc & Infectious Disease Research Corp., Boynton Beach, Florida
  - Daniel A. Warner/Consultive Medicine, Daytona Beach, Florida
  - The McGregor Clinic, Fort Myers, Florida
  - Associates in Infectious Disease, Ft. Pierce, Florida
  - Duval County Health Department, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Care Resource, Miami, Florida
  - South Florida Infectious Deisease and Tropical Medicine Center, Miami, Florida
  - Office of Albert Canas, MD, Miami Beach, Florida
  - Health Positive, Safety Harbor, Florida
  - Pinellas Care Clinic, St. Petersburg, Florida
  - Infectious Disease Research Institute, Inc, Tampa, Florida
  - Midtown Medical Center, Tampa, Florida
  - St. Joseph's Hospital Comprehensive Research Institute, Tampa, Florida
  - Tampa Care Clinic, Tampa, Florida
  - Rowan Tree Medical, PA, Wilton Manors, Florida
  - Atlanta Infectious Disease Group, Atlanta, Georgia
  - Atlanta Primary Care, Atlanta, Georgia
  - PMI Health Research Group, Atlanta, Georgia
  - Family Health Care of Atlanta, PC, Atlanta, Georgia
  - Absolute Care Medical Center, Atlanta, Georgia
  - Kaiser Permanente, Atlanta, Georgia
  - Atlanta Specialty Research, Atlanta, Georgia
  - Georgia Health Sciences University, Augusta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - WellStar Clinical Trials Office, Marietta, Georgia
  - WellStar Infectious Disease, Marietta, Georgia
  - WellStar Kennestone Hospital, Marietta, Georgia
  - Infectious Diseases Associates, Riverdale, Georgia
  - Chatham County Health Department, Savannah, Georgia
  - Ruth M. Rothstein CORE Center, Chicago, Illinois
  - Howard Brown Health Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Office of William Johnson, M.D., Olympia Fields, Illinois
  - Southside Health Association, Olympia Fields, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Blue Grass Care Clinic, Lexington, Kentucky
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - Montgomery Infectious Disease Associates, P.A. (Private Practice), Silver Spring, Maryland
  - St. Elizabeth's Medical Center, Brighton, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - Baystate Infectious Diseases Clinical Research, Springfield, Massachusetts
  - University Of Michigan Health Systems, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St. John hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Ingham County Health Department, Lansing, Michigan
  - Michigan State University College of Osteopathic Medicine, Lansing, Michigan
  - Newland Medical Associates, Southfield, Michigan
  - Federal Medical Center Rochester, Rochester, Minnesota
  - Mayo Medical Clinic, Rochester, Minnesota
  - Nemechek Health Renewal, Kansas City, Missouri
  - Central West Clinical Research, St Louis, Missouri
  - Monmouth Medical Center, Long Branch, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Meridian Medical Associates, Neptune City, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - Erie County Medical Center, HIV Services, Buffalo, New York
  - Guthrie Medical Group, Ithaca, New York
  - North Shore University Hospital, Manhasset, New York
  - Beth Israel Medical Center, New York, New York
  - Beth Israel Medical Clinic, New York, New York
  - Mount Sinai Beth Israel Medical Center, New York, New York
  - HIV & Internal Medicine, New York, New York
  - Mount Sinai Downtown Comprehensive Health Program, New York, New York
  - Columbia University Medical Center, New York, New York
  - CUMC Research Pharmacy, New York, New York
  - AIDS Care, Rochester, New York
  - New York Medical College, Valhalla, New York
  - Westchester Medical Center, Valhalla, New York
  - ID Associates, Gastonia, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Rosedale Infectious Diseases, Huntersville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - University of Toledo: Health Sciences Campus, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - The Research and Education Group, Portland, Oregon
  - Kaiser Permanente Northwest Region, Immune Deficiency Clinic, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Pinnacle Health Medical Services, Harrisburg, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Philadelphia Fight, Philadelphia, Pennsylvania
  - Guthrie Clinic, Ltd., Sayre, Pennsylvania
  - Low Country Infectious Diseases, P.A., Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - MCC Clinic, Columbia, South Carolina
  - University of South Carolina School of Medicine, Columbia, South Carolina
  - University Speciality Clinics, Columbia, South Carolina
  - Central Texas Clinical Research, Austin, Texas
  - Saint Hope Foundation, Bellaire, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - Southwest Infectious Disease Clinical Research, Inc., Dallas, Texas
  - UT Southwestern Medical Center HIV/AIDS Research Unit, Dallas, Texas
  - Pillar Clinical Research LLC, Dallas, Texas
  - Office of Allan Rowan Kelly MD, Fort Worth, Texas
  - Tarrant County Infectious Disease Assocciates, Fort Worth, Texas
  - Tarrant County Infectious Disease Associates, Fort Worth, Texas
  - Garcias' Family Health Group, Harlingen, Texas
  - Valley Aids Council, Harlingen, Texas
  - Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas
  - Diversified Medical Practices, PA, Houston, Texas
  - Dr. Howard Kussman, MD, Plano, Texas
  - University Health Care System, San Antonio, Texas
  - South Texas Veterans Health Care System, San Antonio, Texas
  - Infectious Diseases Associates of Central Virginia, Danville, Virginia
  - Infectious Diseases Associates of Central Virginia, Lynchburg, Virginia
  - Group Health Cooperative, Seattle, Washington
  - Marshall University Joan C. Edwards School of Medicine, Huntington, West Virginia
- Belgium (5):
  - Institute of Tropical Medicine, Antwerp
  - CHU Saint Pierre, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gasthuisberg, Inwendige Geneeskunde, Leuven
  - C.H.U. Sart-Tilman, Liège
- Brazil (6):
  - Hospital Dia, Brasília, Federal District
  - Instituto A.Z. de Pesquisa e Ensino, Curitiba, Paraná
  - Hospital Geral de Nova Iguacu, Nova Iguaçu, Rio de Janeiro
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Centro de Referencia e Treinamento DST/AIDS, São Paulo, São Paulo
  - Hospital Heliopolis, São Paulo, São Paulo
- Canada (7):
  - University of British Columbia/ Downtown Infectious Diseases Clinic, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Clinique Medicale du Quartier Latin, Montreal, Quebec
  - CHUM, Hotel-Dieu Hospital, Montreal, Quebec
  - Recherche Clinique Médicale des Campus, Québec, Quebec
- France (15):
  - Hopital Jean Verdier, Unite de maladies infectieuses, Bondy
  - Hopital Saint-andre CHU de Bordeaux, Bordeaux
  - Hopital Pellegrin, Bordeaux
  - Raymond Poincare Hospital, Garches
  - Hopital de L'Hotel Dieu, Lyon
  - Hopital Sainte Marguerite, Marseille
  - Saint-Louis Hospital, Paris
  - Cochin Hospital Saint Vincent de Paul, Paris
  - Hopital Tenon, Paris
  - Hopital Pitie Salpetriere, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - CH Perpignan, Perpignan
  - Hôpital Haut - Leveque - Centre Francois Magendie, Pessac
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Centre Hospitalier de Tourcoing, Tourcoing
- Germany (20):
  - Arztpraxis fuer Innere Medizin Dr. Knechten, Aachen
  - Praxis City Ost Medizinisches Zentrum, Berlin
  - Praxis Dr. Christiane Cordes, Berlin
  - Klinik I fuer Innere Medizin der Uni-Klinik Koeln, Cologne
  - Klinikum Dortmund, Dortmund
  - Universitaetsklinikum Carl Gustav Carus, Klinik und Poliklinik fuer Dermatologie, Dresden
  - Hospital of the J.W. Goethe University, Medical Clinic II, Frankfurt am Main
  - Praxis Dr. Lothar Schneider Interne Medizin, HIV Schwerpunkt, Fürth
  - IPM - Study - Center, Hamburg
  - ifi-Institut am Allgemeines Krankenhaus St.Georg, Hamburg
  - Universitaetsklinikum Hamburg-Eppendorf, Ambulanzzentrum des UKE GmbH, Bereich Infektiologie, Hamburg
  - Universitaetsklinikum Mainz, I. Medizinische Klinik und Poliklinik,, Mainz
  - Mannheimer Onkologie Praxis, Mannheim
  - Gemeinschaftspraxis Untersendling, München
  - Medizinisches Versorgungszentrum, München
  - Ludwig-Maximilians-Universitaet, Klinikum Innenstadt, Medizinische Poliklinik, München
  - Centrum fuer interdisziplinaere Medizin Muenster GmbH, Münster
  - Klinikum Osnabruck, Osnabrück
  - Infectomed GbR Zentrum für medizinische Studien, Stuttgart
  - Privatpraxis Ulmer, Frietsch, Müller, Stuttgart
- Greece (3):
  - University Hospital of Patras, Pátrai, Achaia
  - Andreas Syngros Hospital, Athens
  - Tzaneion General Hospital of Piraeus, Piraeus
- Italy (23):
  - Clinica Malattie Infettive, Bari
  - Ambulatorio Day Hospital Malattie Infettive, Bologna
  - Dipartimento di Medicina Clinica Specialistica e Sperimentale, Bologna
  - Busto Arsizio Hospital, Busto Arsizio
  - SOD Malattie Infettive, La Piastra dei Servizi, Florence
  - Ente Ospedaliero Ospedali Galliera, Genova
  - San Raffaele Hospital, Milan
  - Clinic of Infectious and Tropical Diseases-University of Milan-San Paolo Hospital, Milan
  - 1 Divisione di Malattive Infettive e Servizio di Allergologia, Ospedale L. Sacco, Milan
  - Universita' degli Studi di Milano, Dipartimento di scienza clinica Luigi Sacco, Milan
  - Azienda Ospedaliero Universitaria Policlinico di Modena, Modena
  - Azienda Ospedal Universitaria II Univ degli Studi di Napoli Servizio di Diagnosi e Terapia, Naples
  - Azienda Ospedaliera "Domenico Cotugno", Napoli
  - AOUP Paolo Giaccone, UOC Malattie Infettive, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Sanitaria Locale Ospedale Civile dello Spirito Santo Presidio Ospedaliero, Pescara
  - Istituto Nazionale Malattie Infettive "L.Spallanzani"-IRCCS, Roma
  - Istituto Nazionale Malattie Infettive INMI- "L. Spallanzani"- I.R.C.C.S., Roma
  - Universita' di Roma La Sapienza, Dipartimento di Malattie Infettive e Tropicali, Roma
  - Universita'Cattolica del Sacro Cuore Policlinico Gemelli, Roma
  - Azienda Ospedaliera San Giovanni Addolorata Presidia Santa Maria, Rome
  - Ospedale Amedeo di Savoia, Torino
  - Ospedale Amedeo di Savoia, Clinica Universitaria di Malattie Infettive, Torino
- Puerto Rico (2):
  - Ararat Research Center, Ponce, PR
  - HOPE Clinical Research, San Juan
- Spain (26):
  - Clinica Mutua de Terrassa, Terrassa, Barcelona
  - Hospital San Pedro, Logroño, La Rioja
  - Hospital de Tortosa Verge de La Cinta, Tortosa, Tarragona
  - Complejo Hospitalario Juan Canalejo, A Coruña
  - Hospital General Universitário de Alicante, Alicante
  - Hospital Del Mar, Barcelona
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital Universitario Germans Tias I Pujol, Barcelona
  - Unidad de Enfermedades Infecciosas, Cadiz
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Donostia, Donostia / San Sebastian
  - Hospital General Universitario de Elche, Elche
  - Hospital Clinico San Cecilio, Granada
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Carlos Iii, Madrid
  - Hospital Ramon Y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Univ. La Paz, Madrid
  - Hospital de Mostoles, Madrid
  - Mataro Hospital, Mataró
  - Complejo Hospitalario Carlos Haya, Málaga
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Virgen de La Macarena, Seville
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Clinico Universitario, Valencia
- United Kingdom (17):
  - Hull & East Yorkshire Hospitals NHS Trust, Cottingham, EAST Yorkshire
  - Clinical Resource Building, Level 7, Newcastle upon Tyne, Newcastle
  - Royal Victoria Hospital, Belfast
  - Selly Oak Hospital, Birmingham
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - North Manchester General Hospital, Crumpsall
  - Darlington Memorial Hospital, Darlington
  - Regional Infectious Diseases Unit, Edinburgh
  - Grahame Hayton Unit, London
  - North Middlesex Hospital, London
  - Royal Free Hospital, Ian Charleson Day Centre, London
  - 1st Floor St Stephens Centre, London
  - Royal Victoria Infirmary Hospital, Newcastle upon Tyne
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Warren browne Unit, Southlands Hospital, Shoreham-by-Sea
  - Cobridge Community Health Centre, Stoke-on-Trent
  - St. George's Hospital, Tooting

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was conducted at multiple sites between 31 March 2008 and 14 February 2019.
Groups:
- Maraviroc Exposed: Human immunodeficiency virus- 1( HIV-1) infected, treatment-experienced adult participants, who were prescribed with maraviroc along with an optimized background antiretroviral therapy (OBT) regimen (in usual clinical practice following the approved local label of maraviroc), were included in this study and were observed in this study for an observation period of up to 5 years following enrollment.
- Maraviroc Unexposed: HIV-1 infected, treatment-experienced adult participants, who were not prescribed with maraviroc but with OBT regimen (in usual clinical practice following the approved local label of maraviroc), were included in this study and were observed in this study for an observation period of up to 5 years following enrollment.
Period: Overall Study
Arm/Group | Maraviroc Exposed | Maraviroc Unexposed
Started | 1316 | 1130
Completed | 814 | 596
Not Completed | 502 | 534
Not completed — Death recorded on subject summary pages | 75 | 75
Not completed — Does not meet entrance criteria | 19 | 21
Not completed — Lost to Follow-up | 203 | 264
Not completed — Withdrawal by Subject | 74 | 65
Not completed — Other | 123 | 108
Not completed — Site closed | 8 | 0
Not completed — Withdrawn due to pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set: All participants who were enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Maraviroc Exposed | Maraviroc Unexposed | Total
Number analyzed (Participants) | 1316 | 1130 | 2446
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (9.3) | 44.3 (10.0) | 45.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 275 | 265 | 540
  Male | 1041 | 865 | 1906
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 983 | 684 | 1667
  Black | 271 | 390 | 661
  Asian | 13 | 7 | 20
  Other | 48 | 48 | 96
  Unspecified | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Density Rate Per 1000 Participant-Years for Incidence of Centers for Disease Control and Prevention Category C AIDS -Defining Opportunistic Infections
Description: Density rate per 1000 participant-years for incidence of centers for disease control and prevention category C acquired immunodeficiency syndrome (AIDS) -defining opportunistic infections was reported. Density rate was calculated as the number of events (n) per 1000 participant-years at risk. Poisson regressions were fit to the categorical events with only treatment in the model to obtain the crude rate and confidence interval (CI).
Time Frame: Up to 5 years following enrollment
Population: Safety analysis set included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: events per 1000 participant-years
Arm/Group | Maraviroc Exposed | Maraviroc Unexposed
Number analyzed (Participants) | 1316 | 1130
events per 1000 participant-years | 22.28 [18.57 to 26.73] | 41.77 [36.09 to 48.34]
Statistical Analysis 1: Comparison: Maraviroc Exposed vs Maraviroc Unexposed; Poisson regressions were fit to the categorical events with only treatment in the model to obtain the crude risk ratio (RR) and CI; Test type: Superiority; Risk Ratio (RR) = 0.53, 95% CI 2-sided [0.42 to 0.67]

2. Primary Outcome: Density Rate Per 1000 Participant-Years for Incidence of Viral Encephalitis
Description: Density rate per 1000 participant-years for incidence of viral encephalitis was reported. Density rate was calculated as the number of events (n) per 1000 participant-years at risk. Poisson regressions were fit to the categorical events with only treatment in the model to obtain the crude rate and CI.
Time Frame: Up to 5 years following enrollment
Population: Safety analysis set included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: events per 1000 participant-years
Arm/Group | Maraviroc Exposed | Maraviroc Unexposed
Number analyzed (Participants) | 1316 | 1130
events per 1000 participant-years | 0.38 [0.10 to 1.54] | 0.46 [0.12 to 1.86]
Statistical Analysis 1: Comparison: Maraviroc Exposed vs Maraviroc Unexposed; Poisson regressions were fit to the categorical events with only treatment in the model to obtain the crude RR and CI; Test type: Superiority; Risk Ratio (RR) = 0.83, 95% CI 2-sided [0.12 to 5.88]

3. Primary Outcome: Density Rate Per 1000 Participant-Years for Incidence of All Malignancies (AIDS Defining Malignancies and Non-AIDS Defining Malignancies)
Description: Density rate per 1000 participant-years for incidence of all malignancies as well as its types (categorized as: AIDS defining malignancies and non-AIDS defining malignancies) were reported. AIDS defining malignancies included malignancies due to any of these: cervical cancer, Kaposi's sarcoma or lymphoma; whereas all other malignancies (except AIDS-defining) were non-aids defining malignancies. Density rate was calculated as the number of events (n) per 1000 participant-years at risk. Poisson regressions were fit to the categorical events with only treatment in the model to obtain the crude rate and CI.
Time Frame: Up to 5 years following enrollment
Population: Safety analysis set included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: events per 1000 participant-years
Arm/Group | Maraviroc Exposed | Maraviroc Unexposed
Number analyzed (Participants) | 1316 | 1130
events per 1000 participant-years
  All Malignancies | 12.87 [10.13 to 16.35] | 13.69 [10.61 to 17.67]
  AIDS defining Malignancies | 2.31 [1.31 to 4.06] | 3.71 [2.27 to 6.06]
  Non-AIDS defining Malignancies | 10.56 [8.11 to 13.76] | 9.98 [7.40 to 13.45]
Statistical Analysis 1: Comparison: Maraviroc Exposed vs Maraviroc Unexposed; All Malignancies: Poisson regressions were fit to the categorical events with only treatment in the model to obtain the crude RR and CI; Test type: Superiority; Risk Ratio (RR) = 0.94, 95% CI 2-sided [0.66 to 1.33]
Statistical Analysis 2: Comparison: Maraviroc Exposed vs Maraviroc Unexposed; AIDS defining Malignancies: Poisson regressions were fit to the categorical events with only treatment in the model to obtain the crude RR and CI; Test type: Superiority; Risk Ratio (RR) = 0.62, 95% CI 2-sided [0.29 to 1.31]
Statistical Analysis 3: Comparison: Maraviroc Exposed vs Maraviroc Unexposed; Non-AIDS defining Malignancies: Poisson regressions were fit to the categorical events with only treatment in the model to obtain the crude RR and CI; Test type: Superiority; Risk Ratio (RR) = 1.06, 95% CI 2-sided [0.71 to 1.58]

4. Primary Outcome: Density Rate Per 1000 Participant-Years for Incidence of Liver Failure
Description: Density rate per 1000 participant-years for incidence of liver failure was reported. Density rate was calculated as the number of events (n) per 1000 participant-years at risk. Poisson regressions were fit to the categorical events with only treatment in the model to obtain the crude rate and CI.
Time Frame: Up to 5 years following enrollment
Population: Safety analysis set included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: events per 1000 participant-years
Arm/Group | Maraviroc Exposed | Maraviroc Unexposed
Number analyzed (Participants) | 1316 | 1130
events per 1000 participant-years | 2.50 [1.45 to 4.30] | 2.55 [1.41 to 4.61]
Statistical Analysis 1: Comparison: Maraviroc Exposed vs Maraviroc Unexposed; Poisson regressions were fit to the categorical events with only treatment in the model to obtain the crude RR and CI; Test type: Superiority; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.44 to 2.18]

5. Primary Outcome: Density Rate Per 1000 Participant-Years for Incidence of Myocardial Infarction or Ischemia: Events Adjudicated as 'Definite' or 'Possible'
Description: Density rate per 1000 participant-years for incidence of myocardial infarction or ischemia (definite + possible) was reported. Events of myocardial infarction or ischemia were adjudicated as definite or possible; where definite= an event had definitely occurred; possible =an event had possibly occurred. Density rate was calculated as the number of events (n) per 1000 participant-years at risk. Poisson regressions were fit to the categorical events with only treatment in the model to obtain the crude rate and CI. In this outcome measure, density rate per 1000 participant-years for incidence of myocardial infarction or ischemia (which included sum of definite + possible events) was reported.
Time Frame: Up to 5 years following enrollment
Population: Safety analysis set included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: events per 1000 participant-years
Arm/Group | Maraviroc Exposed | Maraviroc Unexposed
Number analyzed (Participants) | 1316 | 1130
events per 1000 participant-years | 4.80 [3.24 to 7.11] | 5.34 [3.55 to 8.03]
Statistical Analysis 1: Comparison: Maraviroc Exposed vs Maraviroc Unexposed; Poisson regressions were fit to the categorical events with only treatment in the model to obtain the crude RR and CI; Test type: Superiority; Risk Ratio (RR) = 0.90, 95% CI 2-sided [0.51 to 1.59]

6. Primary Outcome: Density Rate Per 1000 Participant-Years for Incidence of Myocardial Infarction or Ischemia: Events Adjudicated as 'Definite' or 'Possible' or 'Insufficient Data'
Description: Density rate per 1000 participant-years for incidence of myocardial infarction or ischemia (definite + possible + insufficient data) was reported. Events of myocardial infarction or ischemia were adjudicated as definite or possible or insufficient data; where definite= an event had definitely occurred; possible =an event had possibly occurred; insufficient =insufficient data to determine whether an event had occurred. Density rate was calculated as the number of events (n) per 1000 participant-years at risk. Poisson regressions were fit to the categorical events with only treatment in the model to obtain the crude rate and CI. In this outcome measure, density rate per 1000 participant-years for incidence of myocardial infarction or ischemia (which included sum of definite + possible events + insufficient data) was reported.
Time Frame: Up to 5 years following enrollment
Population: Safety analysis set included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: events per 1000 participant-years
Arm/Group | Maraviroc Exposed | Maraviroc Unexposed
Number analyzed (Participants) | 1316 | 1130
events per 1000 participant-years | 8.26 [6.13 to 11.14] | 7.43 [5.25 to 10.50]
Statistical Analysis 1: Comparison: Maraviroc Exposed vs Maraviroc Unexposed; Poisson regressions were fit to the categorical events with only treatment in the model to obtain the crude RR and CI; Test type: Superiority; Risk Ratio (RR) = 1.11, 95% CI 2-sided [0.70 to 1.76]

7. Primary Outcome: Density Rate Per 1000 Participant-Years for Incidence of Rhabdomyolysis
Description: Density rate per 1000 participant-years for incidence of rhabdomyolysis was reported. Density rate was calculated as the number of events (n) per 1000 participant-years at risk. Poisson regressions were fit to the categorical events with only treatment in the model to obtain the crude rate and CI.
Time Frame: Up to 5 years following enrollment
Population: Safety analysis set included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: events per 1000 participant-years
Arm/Group | Maraviroc Exposed | Maraviroc Unexposed
Number analyzed (Participants) | 1316 | 1130
events per 1000 participant-years | 0.77 [0.29 to 2.05] | 0.70 [0.22 to 2.16]
Statistical Analysis 1: Comparison: Maraviroc Exposed vs Maraviroc Unexposed; Poisson regressions were fit to the categorical events with only treatment in the model to obtain the crude RR and CI; Test type: Superiority; Risk Ratio (RR) = 1.10, 95% CI 2-sided [0.25 to 4.93]

8. Primary Outcome: Density Rate Per 1000 Participant-Years for Incidence of Death From Liver-Related Cause
Description: Density rate per 1000 participant-years for incidence of death from liver-related cause was reported. Density rate was calculated as the number of events (n) per 1000 participant-years at risk. Poisson regressions were fit to the categorical events with only treatment in the model to obtain the crude rate and CI.
Time Frame: Up to 5 years following enrollment
Population: Safety analysis set included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: events per 1000 participant-years
Arm/Group | Maraviroc Exposed | Maraviroc Unexposed
Number analyzed (Participants) | 1316 | 1130
events per 1000 participant-years | 0.77 [0.29 to 2.05] | 1.16 [0.48 to 2.79]
Statistical Analysis 1: Comparison: Maraviroc Exposed vs Maraviroc Unexposed; Poisson regressions were fit to the categorical events with only treatment in the model to obtain the crude RR and CI; Test type: Superiority; Risk Ratio (RR) = 0.66, 95% CI 2-sided [0.18 to 2.47]

9. Primary Outcome: Density Rate Per 1000 Participant-Years for Incidence of Death Due to Any Cause
Description: Density rate per 1000 participant-years for incidence of death due to any cause was reported. Density rate was calculated as the number of events (n) per 1000 participant-years at risk. Poisson regressions were fit to the categorical events with only treatment in the model to obtain the crude rate and CI.
Time Frame: Up to 5 years following enrollment
Population: Safety analysis set included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: events per 1000 participant-years
Arm/Group | Maraviroc Exposed | Maraviroc Unexposed
Number analyzed (Participants) | 1316 | 1130
events per 1000 participant-years | 14.41 [11.49 to 18.07] | 18.33 [14.70 to 22.86]
Statistical Analysis 1: Comparison: Maraviroc Exposed vs Maraviroc Unexposed; Poisson regressions were fit to the categorical events with only treatment in the model to obtain the crude RR and CI; Test type: Superiority; Risk Ratio (RR) = 0.79, 95% CI 2-sided [0.57 to 1.08]

10. Primary Outcome: Adjusted Density Rate Per 1000 Participant-Years for Incidence of Centers for Disease Control and Prevention Category C Aids-Defining Opportunistic Infections
Description: Adjusted density rate per 1000 participant-years for incidence of centers for disease control and prevention category c aids-defining opportunistic infections was reported. Density rate was calculated as the number of events (n) per 1000 participant-years at risk. Poisson regressions were fit to the categorical events with treatment as the main effect, propensity score (PS) quartile and imputed Framingham score (FS) as covariates in the model to obtain the adjusted rate and CI.
Time Frame: Up to 5 years following enrollment
Population: Safety analysis set included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: events per 1000 participant-years
Arm/Group | Maraviroc Exposed | Maraviroc Unexposed
Number analyzed (Participants) | 1316 | 1130
events per 1000 participant-years | 22.36 [18.56 to 26.94] | 28.70 [23.98 to 34.34]
Statistical Analysis 1: Comparison: Maraviroc Exposed vs Maraviroc Unexposed; Poisson regressions were fit to the categorical events with treatment as the main effect, PS quartile and imputed FS as covariates in the model to obtain the adjusted RR and CI; Test type: Superiority; Risk Ratio (RR) = 0.78, 95% CI 2-sided [0.61 to 0.99]

11. Primary Outcome: Adjusted Density Rate Per 1000 Participant-Years for Incidence of All Malignancies (AIDS Defining Malignancies and Non-AIDS Defining Malignancies)
Description: Adjusted density rate per 1000 participant-years for incidence of all malignancies as well as its types (categorized as AIDS defining malignancies and non-AIDS defining malignancies) were reported. AIDS defining malignancies included malignancies due to any of these: cervical cancer, Kaposi's sarcoma or lymphoma; whereas all other malignancies (except AIDS-defining) were non-AIDS defining malignancies. Density rate was calculated as the number of events (n) per 1000 participant-years at risk. Poisson regressions were fit to the categorical events with treatment as the main effect, PS quartile and imputed FS as covariates in the model to obtain the adjusted rate and CI.
Time Frame: Up to 5 years following enrollment
Population: Safety analysis set included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: events per 1000 participant-years
Arm/Group | Maraviroc Exposed | Maraviroc Unexposed
Number analyzed (Participants) | 1316 | 1130
events per 1000 participant-years
  All Malignancies | 12.49 [9.72 to 16.05] | 13.54 [10.44 to 17.56]
  AIDS defining Malignancies | 2.31 [1.29 to 4.13] | 3.31 [1.95 to 5.62]
  Non-AIDS defining Malignancies | 9.87 [7.44 to 13.09] | 9.86 [7.27 to 13.37]
Statistical Analysis 1: Comparison: Maraviroc Exposed vs Maraviroc Unexposed; All malignancies: Poisson regressions were fit to the categorical events with treatment as the main effect, PS quartile and imputed FS as covariates in the model to obtain the adjusted RR and CI; Test type: Superiority; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.64 to 1.33]
Statistical Analysis 2: Comparison: Maraviroc Exposed vs Maraviroc Unexposed; AIDS defining malignancies: Poisson regressions were fit to the categorical events with treatment as the main effect, PS quartile and imputed FS as covariates in the model to obtain the adjusted RR and CI; Test type: Superiority; Risk Ratio (RR) = 0.70, 95% CI 2-sided [0.32 to 1.52]
Statistical Analysis 3: Comparison: Maraviroc Exposed vs Maraviroc Unexposed; Non-AIDS defining malignancies: Poisson regressions were fit to the categorical events with treatment as the main effect, PS quartile and imputed FS as covariates in the model to obtain the adjusted RR and CI; Test type: Superiority; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.66 to 1.52]

12. Primary Outcome: Adjusted Density Rate Per 1000 Participant-Years for Incidence of Myocardial Infarction or Ischemia: Events Adjudicated as 'Definite' or 'Possible'
Description: Adjusted density rate per 1000 participant-years for incidence of myocardial infarction or ischemia (definite + possible) was reported. Events of myocardial infarction or ischemia were adjudicated as definite or possible; where definite= an event had definitely occurred; possible =an event had possibly occurred. Density rate was calculated as the number of events (n) per 1000 participant-years at risk. Poisson regressions were fit to the categorical events with treatment as the main effect, PS quartile and imputed FS as covariates in the model to obtain the adjusted rate and CI. In this outcome measure, adjusted density rate per 1000 participant-years for incidence of myocardial infarction or ischemia (which included sum of definite + possible events) was reported.
Time Frame: Up to 5 years following enrollment
Population: Safety analysis set included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: events per 1000 participant-years
Arm/Group | Maraviroc Exposed | Maraviroc Unexposed
Number analyzed (Participants) | 1316 | 1130
events per 1000 participant-years | 2.08 [1.21 to 3.56] | 3.37 [2.06 to 5.52]
Statistical Analysis 1: Comparison: Maraviroc Exposed vs Maraviroc Unexposed; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.62, 95% CI 2-sided [0.35 to 1.10]

13. Primary Outcome: Adjusted Density Rate Per 1000 Participant-Years for Incidence of Myocardial Infarction or Ischemia: Events Adjudicated as 'Definite' or 'Possible' or 'Insufficient Data'
Description: Adjusted density rate per 1000 participant-years for incidence of myocardial infarction or ischemia (definite + possible + insufficient data) was reported. Events of myocardial infarction or ischemia were adjudicated as definite or possible or insufficient data; where definite= an event had definitely occurred; possible =an event had possibly occurred; insufficient =insufficient data to determine whether an event had occurred. Density rate was calculated as the number of events (n) per 1000 participant-years at risk. Poisson regressions were fit to the categorical events with treatment as the main effect, PS quartile and imputed FS as covariates in the model to obtain the adjusted rate and CI. In this outcome measure, adjusted density rate per 1000 participant-years for incidence of myocardial infarction or ischemia (which included sum of definite + possible events + insufficient data) was reported.
Time Frame: Up to 5 years following enrollment
Population: Safety analysis set included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: events per 1000 participant-years
Arm/Group | Maraviroc Exposed | Maraviroc Unexposed
Number analyzed (Participants) | 1316 | 1130
events per 1000 participant-years | 5.65 [3.97 to 8.05] | 5.99 [4.13 to 8.68]
Statistical Analysis 1: Comparison: Maraviroc Exposed vs Maraviroc Unexposed; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.94, 95% CI 2-sided [0.59 to 1.52]

14. Primary Outcome: Adjusted Density Rate Per 1000 Participant-Years for Incidence of Death Due to Any Cause
Description: Adjusted density rate per 1000 participant-years for incidence of death due to any cause was reported. Density rate was calculated as the number of events (n) per 1000 participant-years at risk. Poisson regressions were fit to the categorical events with treatment as the main effect, PS quartile and imputed FS as covariates in the model to obtain the adjusted rate and CI.
Time Frame: Up to 5 years following enrollment
Population: Safety analysis set included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: events per 1000 participant-years
Arm/Group | Maraviroc Exposed | Maraviroc Unexposed
Number analyzed (Participants) | 1316 | 1130
events per 1000 participant-years | 14.39 [11.41 to 18.16] | 15.64 [12.30 to 19.89]
Statistical Analysis 1: Comparison: Maraviroc Exposed vs Maraviroc Unexposed; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.66 to 1.28]

15. Primary Outcome: Percentage of Participants With All-Cause Mortality
Description: All-cause death was defined as the death due to any cause during the course of study.
Time Frame: Up to 5 years following enrollment
Population: Safety analysis set included all participants who were enrolled in the study.
Measure: Number; unit: Percentage of participants
Arm/Group | Maraviroc Exposed | Maraviroc Unexposed
Number analyzed (Participants) | 1316 | 1130
Percentage of participants | 5.7 | 7.0
Statistical Analysis 1: Comparison: Maraviroc Exposed vs Maraviroc Unexposed; Test type: Superiority; p = 0.6225, Regression, Cox; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.66 to 1.28]

ADVERSE EVENTS:
Time Frame: Up to 5 years following enrollment
Description: Same event may appear as adverse event (AE) and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another or 1 participant may have experienced both serious and non-serious event during study. Four participants in the arm "MVC-unexposed group" were not counted under "death" reason of discontinuation, because these deaths were not recorded on participant summary page at the time of "reason of discontinuation" analysis.
Arm/Group | Maraviroc Exposed | Maraviroc Unexposed
All-Cause Mortality (participants affected / at risk) | 75/1316 | 79/1130
Serious Adverse Events (participants affected / at risk) | 435/1316 | 352/1130
Other Adverse Events (participants affected / at risk) | 111/1316 | 34/1130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Maraviroc Exposed (N=1316) | Maraviroc Unexposed (N=1130)
Anaemia (Blood and lymphatic system disorders) | 11 | 14
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 2
Haemolysis (Blood and lymphatic system disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 2 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 2
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 1
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 2
Pancytopenia (Blood and lymphatic system disorders) | 3 | 5
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 7 | 6
Angina pectoris (Cardiac disorders) | 2 | 1
Angina unstable (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 6
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 5 | 2
Cardiac failure (Cardiac disorders) | 4 | 1
Cardiac failure congestive (Cardiac disorders) | 5 | 11
Cardiac valve disease (Cardiac disorders) | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 4 | 1
Cardiogenic shock (Cardiac disorders) | 2 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 2
Congestive cardiomyopathy (Cardiac disorders) | 0 | 2
Coronary artery disease (Cardiac disorders) | 6 | 4
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 2 | 3
Myocardial infarction (Cardiac disorders) | 16 | 12
Myocardial ischaemia (Cardiac disorders) | 3 | 1
Myocarditis (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 1
Torsade de pointes (Cardiac disorders) | 1 | 0
Fanconi syndrome (Congenital, familial and genetic disorders) | 1 | 1
Sickle cell disease (Congenital, familial and genetic disorders) | 0 | 1
Deafness bilateral (Ear and labyrinth disorders) | 0 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 2
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 3 | 1
Adrenal mass (Endocrine disorders) | 1 | 0
Autoimmune hypothyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1
Cataract (Eye disorders) | 4 | 0
Central vision loss (Eye disorders) | 1 | 0
Iridocyclitis (Eye disorders) | 1 | 0
Orbital cyst (Eye disorders) | 0 | 1
Pupils unequal (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 1 | 1
Vision blurred (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 8 | 11
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 1
Anal skin tags (Gastrointestinal disorders) | 1 | 0
Anogenital dysplasia (Gastrointestinal disorders) | 1 | 0
Anorectal disorder (Gastrointestinal disorders) | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 4 | 3
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 5 | 2
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 13
Diverticulum (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 2 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 3
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Haematemesis (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 4 | 2
Intestinal ischaemia (Gastrointestinal disorders) | 2 | 0
Intestinal mass (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Intussusception (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 2 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 2
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal rupture (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 6 | 2
Pancreatitis acute (Gastrointestinal disorders) | 1 | 6
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 2
Proctitis ulcerative (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Rectal perforation (Gastrointestinal disorders) | 1 | 0
Rectal prolapse (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 3
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 4
Asthenia (General disorders) | 1 | 5
Chest pain (General disorders) | 16 | 15
Chills (General disorders) | 0 | 1
Death (General disorders) | 10 | 6
Dysplasia (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 1
Gait disturbance (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 2 | 1
Generalised oedema (General disorders) | 1 | 0
Hypothermia (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Multi-organ disorder (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Physical deconditioning (General disorders) | 1 | 0
Pyrexia (General disorders) | 8 | 11
Sudden cardiac death (General disorders) | 1 | 1
Sudden death (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Treatment noncompliance (General disorders) | 2 | 1
Ulcer (General disorders) | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 1
Biliary dilatation (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 4 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 4 | 2
Hepatic failure (Hepatobiliary disorders) | 3 | 4
Hepatitis alcoholic (Hepatobiliary disorders) | 0 | 2
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Jarisch-Herxheimer reaction (Immune system disorders) | 0 | 1
AIDS related complication (Infections and infestations) | 1 | 0
AIDS retinopathy (Infections and infestations) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal sepsis (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 2 | 1
Abscess limb (Infections and infestations) | 0 | 4
Acquired immunodeficiency syndrome (Infections and infestations) | 2 | 6
Acute hepatitis C (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 2
Amoebiasis (Infections and infestations) | 1 | 2
Amoebic dysentery (Infections and infestations) | 0 | 2
Anal abscess (Infections and infestations) | 0 | 2
Anorectal cellulitis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 7 | 4
Arthritis bacterial (Infections and infestations) | 1 | 2
Aspergillus infection (Infections and infestations) | 0 | 1
Atypical mycobacterial infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 2 | 5
Bacterial diarrhoea (Infections and infestations) | 1 | 1
Bacterial infection (Infections and infestations) | 1 | 0
Brain abscess (Infections and infestations) | 1 | 0
Breast abscess (Infections and infestations) | 0 | 2
Bronchiolitis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 10 | 6
Bronchitis viral (Infections and infestations) | 1 | 0
Burkholderia cepacia complex sepsis (Infections and infestations) | 0 | 1
CNS ventriculitis (Infections and infestations) | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 2 | 0
Campylobacter infection (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 12 | 18
Cellulitis staphylococcal (Infections and infestations) | 0 | 1
Cerebral toxoplasmosis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 3
Clostridium difficile infection (Infections and infestations) | 0 | 4
Corneal abscess (Infections and infestations) | 1 | 0
Cryptococcal fungaemia (Infections and infestations) | 0 | 1
Cryptococcosis (Infections and infestations) | 0 | 1
Cryptosporidiosis infection (Infections and infestations) | 0 | 1
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 | 1
Cytomegalovirus colitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 2
Cytomegalovirus viraemia (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 1 | 1
Device related sepsis (Infections and infestations) | 0 | 1
Diabetic foot infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 0
Empyema (Infections and infestations) | 1 | 1
Encephalitis (Infections and infestations) | 1 | 0
End stage AIDS (Infections and infestations) | 1 | 1
Endocarditis (Infections and infestations) | 1 | 2
Enterococcal sepsis (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 2 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 2
Escherichia urinary tract infection (Infections and infestations) | 0 | 3
External ear cellulitis (Infections and infestations) | 1 | 1
Eye infection syphilitic (Infections and infestations) | 1 | 1
Folliculitis (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Fungal oesophagitis (Infections and infestations) | 1 | 1
Furuncle (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 7 | 11
Gastroenteritis bacterial (Infections and infestations) | 0 | 1
Gastroenteritis clostridial (Infections and infestations) | 1 | 0
Gastroenteritis cryptosporidial (Infections and infestations) | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 2
Genital herpes (Infections and infestations) | 2 | 1
Genital herpes simplex (Infections and infestations) | 1 | 2
Giardiasis (Infections and infestations) | 1 | 0
Gonorrhoea (Infections and infestations) | 1 | 0
HIV enteropathy (Infections and infestations) | 1 | 0
HIV infection (Infections and infestations) | 0 | 2
HIV wasting syndrome (Infections and infestations) | 1 | 2
HIV-associated neurocognitive disorder (Infections and infestations) | 3 | 2
Helicobacter gastritis (Infections and infestations) | 1 | 0
Helicobacter infection (Infections and infestations) | 1 | 2
Hepatitis B reactivation (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 2
Herpes pharyngitis (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 4
Herpes virus infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 5 | 4
Herpes zoster disseminated (Infections and infestations) | 0 | 1
Histoplasmosis (Infections and infestations) | 1 | 2
Infectious colitis (Infections and infestations) | 0 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 4 | 3
Intervertebral discitis (Infections and infestations) | 1 | 0
Joint abscess (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 2
Latent syphilis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 3
Lung infection (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 3 | 1
Meningitis aseptic (Infections and infestations) | 1 | 2
Meningitis cryptococcal (Infections and infestations) | 0 | 4
Meningitis streptococcal (Infections and infestations) | 0 | 1
Meningitis tuberculous (Infections and infestations) | 0 | 1
Microsporidia infection (Infections and infestations) | 0 | 1
Mycobacterial infection (Infections and infestations) | 2 | 0
Mycobacterium abscessus infection (Infections and infestations) | 1 | 0
Mycobacterium avium complex infection (Infections and infestations) | 0 | 4
Mycobacterium fortuitum infection (Infections and infestations) | 0 | 1
Neurosyphilis (Infections and infestations) | 2 | 2
Neutropenic sepsis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 2 | 8
Oral candidiasis (Infections and infestations) | 3 | 3
Oral hairy leukoplakia (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 0 | 2
Osteomyelitis (Infections and infestations) | 1 | 2
Osteomyelitis chronic (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 2
Parvovirus infection (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 3
Peritonitis (Infections and infestations) | 3 | 0
Peritonitis bacterial (Infections and infestations) | 2 | 2
Pharyngitis (Infections and infestations) | 0 | 2
Pilonidal cyst (Infections and infestations) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 2 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 9 | 13
Pneumonia (Infections and infestations) | 51 | 54
Pneumonia bacterial (Infections and infestations) | 1 | 4
Pneumonia influenzal (Infections and infestations) | 0 | 1
Pneumonia legionella (Infections and infestations) | 1 | 0
Pneumonia necrotising (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 2
Pneumonia pseudomonal (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 2 | 1
Pneumonia streptococcal (Infections and infestations) | 1 | 2
Post procedural infection (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 2
Pyelonephritis (Infections and infestations) | 2 | 5
Pyelonephritis acute (Infections and infestations) | 0 | 3
Rectal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 2
Salmonella sepsis (Infections and infestations) | 0 | 1
Secondary syphilis (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 11 | 11
Sepsis syndrome (Infections and infestations) | 0 | 1
Septic embolus (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 5 | 3
Shigella infection (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 3 | 3
Sinusitis bacterial (Infections and infestations) | 0 | 1
Sinusitis fungal (Infections and infestations) | 1 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 3
Staphylococcal infection (Infections and infestations) | 3 | 4
Staphylococcal skin infection (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 4
Superinfection bacterial (Infections and infestations) | 0 | 1
Syphilis (Infections and infestations) | 3 | 1
Syphilis anal (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Toxoplasmosis (Infections and infestations) | 0 | 1
Trichomoniasis (Infections and infestations) | 1 | 1
Tuberculosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 10 | 8
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 2 | 1
Vaginal infection (Infections and infestations) | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Vulval abscess (Infections and infestations) | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1
Accident (Injury, poisoning and procedural complications) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 3 | 1
Breast injury (Injury, poisoning and procedural complications) | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 | 1
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal stoma necrosis (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 2
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 2 | 0
Overdose (Injury, poisoning and procedural complications) | 7 | 3
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Radial nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 3 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Splenic injury (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 3 | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Atypical mycobacterium test positive (Investigations) | 1 | 0
Biopsy lymph gland (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
Body temperature increased (Investigations) | 1 | 0
Culture stool positive (Investigations) | 0 | 1
Drug clearance increased (Investigations) | 1 | 0
Electrocardiogram repolarisation abnormality (Investigations) | 1 | 0
HIV test positive (Investigations) | 0 | 1
Haemophilus test positive (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Liver function test increased (Investigations) | 0 | 1
Staphylococcus test (Investigations) | 1 | 0
Staphylococcus test positive (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 1
Weight decreased (Investigations) | 2 | 1
Alcoholic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 5 | 7
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
Electrolyte depletion (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 2
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 4
Folate deficiency (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Haemochromatosis (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 6
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 4
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 5 | 2
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 3 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Anal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaplastic large cell lymphoma T- and null-cell types (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Diffuse large B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Ocular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Pancreatic carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Plasmablastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Alcoholic seizure (Nervous system disorders) | 1 | 0
Amputation stump pain (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 7 | 4
Clonic convulsion (Nervous system disorders) | 1 | 0
Cranial nerve palsies multiple (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Diabetic hyperglycaemic coma (Nervous system disorders) | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 5
Dysarthria (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 1
Encephalitis post varicella (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 2
Epilepsy (Nervous system disorders) | 1 | 2
Facial paralysis (Nervous system disorders) | 1 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 5
Hemiparesis (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 3 | 5
Hypoaesthesia (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 3 | 0
Lacunar stroke (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Mental impairment (Nervous system disorders) | 0 | 2
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Motor dysfunction (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 2 | 2
Parkinson's disease (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 8 | 5
Somnolence (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 2 | 1
Transient ischaemic attack (Nervous system disorders) | 3 | 0
Unresponsive to stimuli (Nervous system disorders) | 1 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Device dislocation (Product Issues) | 1 | 1
Adjustment disorder (Psychiatric disorders) | 0 | 1
Affective disorder (Psychiatric disorders) | 1 | 0
Aggression (Psychiatric disorders) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 1
Alcoholism (Psychiatric disorders) | 0 | 2
Bipolar I disorder (Psychiatric disorders) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 0
Borderline personality disorder (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 3
Confusional state (Psychiatric disorders) | 2 | 0
Delirium (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 3 | 6
Depression suicidal (Psychiatric disorders) | 0 | 3
Drug abuse (Psychiatric disorders) | 1 | 2
Homicidal ideation (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 1
Mania (Psychiatric disorders) | 1 | 1
Mental status changes (Psychiatric disorders) | 3 | 8
Organic brain syndrome (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 1
Schizoaffective disorder (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 1 | 2
Substance abuse (Psychiatric disorders) | 2 | 2
Substance-induced psychotic disorder (Psychiatric disorders) | 2 | 0
Suicidal ideation (Psychiatric disorders) | 4 | 3
Suicide attempt (Psychiatric disorders) | 4 | 3
Acute kidney injury (Renal and urinary disorders) | 8 | 18
Calculus urinary (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 3
End stage renal disease (Renal and urinary disorders) | 0 | 3
Glomerulonephritis (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 3
Nephropathy (Renal and urinary disorders) | 0 | 2
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 2
Renal failure (Renal and urinary disorders) | 10 | 4
Renal haematoma (Renal and urinary disorders) | 1 | 0
Renal injury (Renal and urinary disorders) | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 1 | 1
Renal vein thrombosis (Renal and urinary disorders) | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Breast enlargement (Reproductive system and breast disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 2
Fallopian tube obstruction (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Ovarian vein thrombosis (Reproductive system and breast disorders) | 1 | 0
Painful erection (Reproductive system and breast disorders) | 0 | 1
Pelvic adhesions (Reproductive system and breast disorders) | 1 | 0
Perineal rash (Reproductive system and breast disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Testicular swelling (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Pulmonary eosinophilia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 1
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 3 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Abdominal hernia repair (Surgical and medical procedures) | 0 | 1
Abscess drainage (Surgical and medical procedures) | 2 | 0
Arterial stent insertion (Surgical and medical procedures) | 1 | 0
Arteriovenous fistula operation (Surgical and medical procedures) | 0 | 1
Cardiac resynchronisation therapy (Surgical and medical procedures) | 1 | 0
Cataract operation (Surgical and medical procedures) | 0 | 1
Colostomy (Surgical and medical procedures) | 1 | 0
Gastric banding reversal (Surgical and medical procedures) | 1 | 0
Hip surgery (Surgical and medical procedures) | 1 | 0
Hysterectomy (Surgical and medical procedures) | 0 | 1
Immune tolerance induction (Surgical and medical procedures) | 0 | 1
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
Leg amputation (Surgical and medical procedures) | 1 | 0
Medical device removal (Surgical and medical procedures) | 0 | 1
Renal transplant (Surgical and medical procedures) | 1 | 0
Valvuloplasty cardiac (Surgical and medical procedures) | 1 | 0
Aortic aneurysm (Vascular disorders) | 2 | 1
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Aortic arteriosclerosis (Vascular disorders) | 1 | 0
Bleeding varicose vein (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 4 | 3
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 6
Hypertensive crisis (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 1 | 7
Hypovolaemic shock (Vascular disorders) | 0 | 1
Iliac artery occlusion (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 3
Peripheral arterial occlusive disease (Vascular disorders) | 3 | 2
Peripheral artery occlusion (Vascular disorders) | 1 | 1
Peripheral artery stenosis (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Subclavian artery thrombosis (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 2 | 0
Thrombosis (Vascular disorders) | 1 | 0
Vascular stenosis (Vascular disorders) | 0 | 1
Vasospasm (Vascular disorders) | 1 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc Exposed (N=1316) | Maraviroc Unexposed (N=1130)
Diarrhoea (Gastrointestinal disorders) | 32 | 14
Nausea (Gastrointestinal disorders) | 18 | 5
Fatigue (General disorders) | 15 | 6
Bronchitis (Infections and infestations) | 18 | 5
Nasopharyngitis (Infections and infestations) | 16 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 3
Headache (Nervous system disorders) | 16 | 6
Rash (Skin and subcutaneous tissue disorders) | 17 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2010-11-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT00665561/Prot_000.pdf
  • Statistical Analysis Plan (2011-03-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT00665561/SAP_001.pdf